CLINICAL TRIAL: NCT06087406
Title: A Phase 1b, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Imvotamab in Participants With Moderate to Severe Rheumatoid Arthritis Who Have Failed Prior Therapies
Brief Title: A Phase 1b Study of Imvotamab in Moderate to Severe Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Interim data from the Phase 1b studies of imvotamab in rheumatoid arthritis demonstrated that the depth and consistency in B Cell depletion required to measure success was insufficient.
Sponsor: IGM Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IGM-2323-102
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis; Arthritis, Rheumatoid; Arthritis
Keywords: Arthritis; Moderate to severe arthritis; active rheumatoid arthritis; bDMARD; tsDMARD; refractory
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imvotamab (Dose Escalation) (Experimental): Imvotatmab administered intravenously
  Interventions: Drug: Imvotamab
- PBO IV (Placebo Comparator): Placebo administered intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imvotamab — Administered intravenously
  Arms: Imvotamab (Dose Escalation)
Drug: Placebo — 0.9% sodium chloride administered intravenously
  Arms: PBO IV

SUMMARY:
The purpose of this study is to determine the safety and tolerability of imvotamab in patients with moderate to severe rheumatoid arthritis who have failed prior therapies.

Participants will be given imvotamab or placebo through a vein (i.e., intravenously). A placebo is a look-alike substance that contains no active drug

DETAILED DESCRIPTION:
This is a Phase 1b, randomized, placebo-controlled, multicenter study to determine the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of imvotamab in adult participants with active RA who are refractory or intolerant to 2 previous biologic disease-modifying anti-rheumatic drugs (bDMARD) or targeted synthetic disease-modifying anti-rheumatic drugs (tsDMARD) therapies. Approximately 40 participants will be sequentially assigned to different dose escalation cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years at the time of signing ICF
* Documented diagnosis of RA and meeting the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for RA at least 1 year prior to screening
* Have had treatment with bDMARDs and/or tsDMARD and were refractory by 1 of 2 reasons:

  * Lack of benefit to at least 2 bDMARDs in different mechanism classes or 1 bDMARD and 1 tsDMARD, after at least 12 weeks of treatment, in the opinion of the investigator. Lack of benefit may include inadequate improvement in joint counts, physical function, or disease activity.
  * Intolerance to at least 2 bDMARDs in different mechanism classes or 1 bDMARD and 1 tsDMARD.
* Minimum of 6 swollen (SJC) and 6 tender joints (TJC) on a 66/68 joint count at the screening and baseline visit (SJC/TJC)
* Central lab results for hsCRP ≥ 0.8 mg/dL
* Anti-citrullinated protein antibodies (ACPA) positive and/or rheumatoid factor (RF) positive
* If using oral corticosteroids (OCS), must be on a stable dose equivalent to ≤ 10 mg/day of prednisone for at least 2 weeks prior to first study treatment

Key Exclusion Criteria:

* History of a rheumatologic autoimmune disease other than RA (except secondary Sjögren's syndrome), or with significant systemic involvement secondary to RA (vasculitis, pulmonary fibrosis, or Felty's syndrome); Juvenile idiopathic arthritis (JIA) or idiopathic arthritis diagnosed before the age of 16 years; Psoriatic Arthritis; Axial spondylarthritis or any other disease associated with inflammatory arthritis; Active fibromyalgia with pain symptoms or signs that would interfere with clinical assessments for RA
* Receipt of an investigational therapy less than 3 months or 5 drug-elimination half-lives (whichever is longer) prior to first administration of study treatment and during the study
* Receipt of any of the following excluded RA therapies:

  * Any cell depleting therapy, anti-CD4, anti-CD5, anti-CD3, rituximab, ocrelizumab, or ofatumumab, less than 6 months prior to first administration of study treatment.
  * Have received prior tsDMARds including but not limited to inhibitors of Janus kinase (JAK), Bruton tyrosine kinase, or tyrosine kinase 2, including baricitinib, tofacitinib, upadacitinib, filgotinib, ibrutinib, or fenebrutinib, or any investigational agent less than 3 months or 5 half-lives, whichever is longer, prior to first administration of study treatment
  * Have received prior immunomodulatory bDMARDs for RA including, but not limited to adalimumab, golimumab, ustekinumab, secukinumab, tocilizumab, abatacept, or other inhibitors of TNF, IL-6, IL-23, or IL-17 less than 3 months or 5 half-lives, whichever is longer, prior to first administration of the study treatment
* Requiring therapy with prednisone > 10 mg/day (or equivalent dose) within 2 weeks prior to first study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of imvotamab in participants with moderate to severe rheumatoid arthritis | Up to Week 52
  Incidence of adverse events (AEs), serious adverse events (SAEs), including serious infectious events (SIEs) and opportunistic infections (OIs)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Humke, MD, Study Director — IGM Biosciences
Locations (18):
- United States (10):
  - Arizona Arthritis & Rheumatology Research, PLLC, Flagstaff, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Glendale, Arizona
  - Triwest Research Associates, San Diego, California
  - East Bay Rheumatology Medical Group, San Leandro, California
  - University of Colorado Hopsital - Anschutz Medical Campus, Aurora, Colorado
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Omega Research MetroWest, Orlando, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - Accelacare - Salisbury, Salisbury, North Carolina
  - Southwest Rheumatology Research, Mesquite, Texas
- Poland (8):
  - Centrum Reumatologii i Rehabilitacji NOVA REUMA, Bialystok, Podlaskie Voivodeship
  - Nova Reuma Domyslawska i Rusilowicz Spólka Partnerska Lekarza Reumatologa i Fizjoterapeuty, Bialystok
  - Medicover Integrated Clinical Services (MCIS) Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Niepubliczny Zakład Opieki Zdrowotnej Lecznica MAK-MED w Nadarzynie, Nadarzyn
  - Med Polonia Sp. z o. o. - Obornicka, Poznan
  - Medyczne Centrum Hetmanska, Poznan
  - Prywatna Praktyka Lekarska Prof. Dr Hab. Med. Paweł Hrycaj, Poznan
  - Reumedika s.c. Wiesława i Łukasz Porawscy, Poznan